CLINICAL TRIAL: NCT00000276
Title: Dopamine Reuptake Inhibitors of Cocaine Abuse
Brief Title: Dopamine Reuptake Inhibitors of Cocaine Abuse - 1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-09250-1; P50DA009250 (NIH); P50-09250-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
The purpose of this study is to evaluate dopamine reuptake inhibitors for cocaine abuse.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-09; Primary Completion 1999-08 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Side effects
Cocaine effects

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States